CLINICAL TRIAL: NCT06009341
Title: The Effect of Pain Management, Relaxation and Fall Training on Clinical Parameters in Total Knee Arthroplasty Patients
Brief Title: Effectiveness of Relaxation Methods in Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Artroplasti gevşeme
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Knee Arthroplasty
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In this study, the intervention group will be given comprehensive training in addition to standard conservative follow-up (pain spasm pain cycle, pain does not always mean that there is a problem, tissue repair, fall prevention, lower extremity classical massage, muscle relaxation relaxation methods, respiratory control), while the control group will be followed only with conservative treatment applications (muscle strengthening, stretching). The applications will be performed with 10 repetitions each day.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will not be trained. Only exercise brochure including muscle strengthening and stretching will be given.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The control group will not be trained. Only exercise brochure including muscle strengthening and stretching will be given. In addition, the intervention group will be taught the training program and applications.

SUMMARY:
In this study, the effectiveness of a comprehensive training program consisting of pain management, relaxation, breathing, massage and falling components will be investigated in patients with total knee arthroplasty. In this randomized controlled study, the trainings will be offered face-to-face after the initial evaluation and within the scope of telemedicine with prepared videos. The first evaluation will be performed on the first postoperative day and the last evaluation will be performed 3 months postoperatively. The aim of this study is to evaluate the effectiveness of a comprehensive education program consisting of pain management, relaxation, respiration, massage and fall components in patients with total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 50 and over
* Participants indicated for unilateral or bilateral total knee arthoplasty
* Individuals to be followed after surgery

Exclusion Criteria:

* Other surgeries
* Individuals with neurological and orthopedic diagnoses
* Individuals with cognitive, hearing, speech and psychiatric problems that prevent them from communicating
* Illiterate individuals
* Presence of malignancy
* Not signing the consent form

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Knee Society Short Form (KSSF) | Change from Baseline KSSF at 12 weeks
  The scale is a 9-item measure developed to assess total knee arthroplasty patients' satisfaction, expectations, physical activities, and clinical and functional status in the preoperative and postoperative period, reported by both the physician and the patient.
Visual Analog Scale (VAS) | Change from Baseline VAS at 12 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 12 weeks
  The questionnaire is a 17-item scale developed to measure fear of movement/reinjury. The normal score range is between 17 and 68.
EQ-5D-3L Quality of Life Scale | Change from Baseline EQ-5D-3L at 12 weeks
  The EQ-5D-3L provides information on three aspects of quality of life. Each dimension has three levels of impairment: no problems (level 1), some problems (level 2) and extreme problems (level 3). The score ranges from less than 0 to 1 (where 0 is a health status equivalent to death and negative values are worse than death) and 1 is the most positive score (the best perceived level according to the five dimensions included in the scale). Finally, the EQ VAS score is obtained by asking patients to rate their health status on a 20 cm vertical scale. The scale ranges from 0 to 100, with 0 meaning "worst imaginable health" and 100 meaning "best imaginable health".
Pain Catastrophising Scale (PCS) | Change from Baseline PCS at 12 weeks
  Scale is used to assess the patient's feelings and thoughts about pain and disaster. The total score ranges from 0 to 52 points. A high score indicates a bad situation.
Activity Specific Balance Confidence Scale (ABC) | Change from Baseline ABC at 12 weeks
  This scale includes 16 tasks related to indoor and outdoor activities of daily living to measure balance confidence in older people with various levels of function. Scores for each question range from 0% (no confidence) to 100% (full confidence). Higher scores indicate greater confidence.
Fear of Falling Avoidance Behavior Questionnaire (FFABQ) | Change from Baseline FFABQ at 12 weeks
  The Fear of Falling Avoidance Behavior Questionnaire (FFABQ) was developed to assess avoidance behavior (activity limitation and participation restriction) in community-dwelling older adults. The FFABQ consists of 14 items ranked using a five-point Likert style, resulting in a maximum possible score of 56 points. A high score indicates activity limitation and participation restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No